CLINICAL TRIAL: NCT04169919
Title: Povidone Iodine 5% Eye Wash in Treatment of Epidemic Keratoconjunctivitis
Brief Title: Modified Treatment for Epidemic Keratoconjunctivitis (EKC)
Acronym: EKC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Shaaban Elwan, Assistant professor of ophthalmology, Minia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Security Forces Hospital, EKC
Record Dates: First submitted 2019-11-13; First posted 2019-11-20 (Actual); Last update posted 2019-11-20 (Actual); Status verified 2019-11

CONDITIONS: Symptoms and Signs
MeSH Terms: conditions — Signs and Symptoms | interventions — Povidone-Iodine

STUDY DESIGN:
Intervention Model Description: Group 1 modified method Group 2 ordinary method
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified method (Active Comparator): Povidone Iodine
  Interventions: Drug: Povidone-Iodine
- Ordinary method (Active Comparator): normal saline
  Interventions: Drug: Normal Saline Flush

INTERVENTIONS:
Drug: Povidone-Iodine — Povidone-Iodine 5% eye wash
  Other Names: Group1
  Arms: Modified method
Drug: Normal Saline Flush — Normal Saline eye wash
  Other Names: Group 2
  Arms: Ordinary method

SUMMARY:
Background: Epidemic Keratoconjunctivitis (EKC) is a form of adenoviral conjunctivitis. It is highly infectious disease mainly affect the outer eye surface and has a frequency to happen in epidemics especially in closed communities such as hospitals, schools and factories.

purpose: The purpose of this study to compare between the modified and the ordinary method of treatment for EKC.

Patients and methods: Three hundred fifty patients of EKC were enrolled in the study. The diagnosis was made by clinical picture and laboratory investigations. Group 1 had two hundred patients 120 males, 80 females (age from 18 to 60 years) were treated by the modified method and group 2 had one hundred fifty patients 100 males,50 females (age from 18 to 58 years) were treated with the ordinary method. The study was hold between November 2014 to October 2018 in Security forces Hospital, Riyadh, Saudi Arabia. Patients were followed up for 3 months up to 2 years. The main outcome were improvement in clinical picture and recovery.

DETAILED DESCRIPTION:
Patients and Methods Three hundred fifty patients suffered from EKC were enrolled in the study. Their diagnosis was made by clinical picture and laboratory investigations. Group 1 had two hundred patients 120 males, 80 females (age from 18 to 60 years) were treated by the modified method and group 2 had one hundred fifty patients 100 males,50 females (age from 18 to 58 years) were treated with the ordinary method. The study was done between November 2014 to October 2018 in Security forces Hospital, Riyadh, Saudi Arabia. Patients were followed up for 3 months up to 2 years. The main outcomes were improvement in patients clinical picture and recovery. All patients signed a consent for inclusion in the study and the study was approved by the ethical committee and it was in agreement with declaration of Helsinki tents.

All cases were diagnosed by clinical symptoms and signs as shown in table (2& 3) and conjunctival smear for some suspected patients which revealed lymphocytes predominance. Slit lamp examination and visual acuity measurement were done and grading of ocular symptoms and signs were estimated according to severerity into normal, mild, moderate or severe. The patients were divided into group 1 in which patients were treated by the modified method (Povidone Iodine 5% eye wash irrigation) and group 2 in which patients were treated by the ordinary method.

Modified method The eye was topically anesthetized, then eye wash with Povidone Iodine 5% (povidone-iodine, Alcon) eye irrigation every day until the patients recovered. Manual removal of pseudo membranes with non toothed forceps and cotton tipped applicator on slit lamp. Antibiotic eye drops (moxifloxacin 0.5%) QID. Lubricant eye drops (tears natural free minims eye drops) QID. Cold compresses. Topical corticosteroid eye drops (fluorometholone 0.1%) QID in cases of subepithelial infiltrates or pseudomemrane formation.

Usual method The same way of management except the eye wash with Povidone Iodine 5% . Steroids was used for symptomatic relief but it do not lower the disease pathway. It suppress the corneal inflammation, improve overall comfort but they also prolong clearance of the virus and the lesions may recur if steroid is prematurely discontinued.

ELIGIBILITY:
Inclusion Criteria:

* Including adult patients with 18 to 60 years old
* Patients with BCDVA of ≥ 20/80 in the study eye
* If the patent have bilateral EKC only one eye included in the study
* Patients attending all the required follow up visits as advised.

Exclusion Criteria:

* Children
* Patients with ocular infection rather than EKC
* Patients with corneal ulceration or bacterial keratitis
* Immunocompromised patients
* Glaucoma
* Patients not attending the required follow up visits.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 350 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Ocular symptoms of epidemic keratoconjunctivitis | 2 weeks
  Ocular symptoms of epidemic keratoconjunctivitis include the following 1-Lid swelling. 2-Red eyes. 3- Watery discharge. 4- Photophobia. 5- Eye discomfort .
  Each symptom evaluated with grade severity:- Normal= no abnormality (0 score), mild= subtle abnormality (1-2 score), moderate= obvious abnormality (3-4 score) and severe = marked abnormality (5 score). the minimum value was 0 score and means better outcome and maximum score is 5 and means worse outcome.
Ocular signs of epidemic keratoconjunctivitis | 2 weeks
  Ocular signs of epidemic keratoconjunctivitis include the following
  1- Lid edema. 2- Follicular conjunctivitis. 3-Pseudomembrane formation. 4- Punctate epithelial keratitis.
  Each sign evaluated with grade severity:- Normal= no abnormality (0 score), mild= subtle abnormality (1-2 score), moderate= obvious abnormality (3-4 score) and severe = marked abnormality (5 score). the minimum value was 0 score and means better outcome and maximum score is 5 and means worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Shaaban A Elwan, MD, Principal Investigator — Minia University and SFH

IPD SHARING:
Plan to Share IPD: Yes
methods
Supporting Information: CSR
Time Frame: 2 years
Access Criteria: Methods and results

REFERENCES:
- [Background] Trinavarat A, Atchaneeyasakul LO. Treatment of epidemic keratoconjunctivitis with 2% povidone-iodine: a pilot study. J Ocul Pharmacol Ther. 2012 Feb;28(1):53-8. doi: 10.1089/jop.2011.0082. Epub 2011 Sep 14. PMID 21916618